CLINICAL TRIAL: NCT03374358
Title: Effect on Liver Fat, Adipose Tissue and Metabolic Parameters When Switching a Protease Inhibitor or Efavirenz to Once Daily Raltegravir in HIV+ Patients With Body Mass Index Over 25 kg/m2 and With at Least One Metabolic Syndrome Component
Brief Title: Effect on Liver Fat and Metabolic Parameters When Switching a Protease Inhibitor or Efavirenz to Raltegravir
Acronym: OBERAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jussi Sutinen, Consultant, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBERAL
Record Dates: First submitted 2017-12-02; First posted 2017-12-15 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: HIV Seropositivity; Metabolic Syndrome; Fatty Liver
MeSH Terms: conditions — HIV Seropositivity; Metabolic Syndrome; Fatty Liver | interventions — Raltegravir Potassium

STUDY DESIGN:
Intervention Model Description: This study is a randomized, open, parallel design study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention arm. (No Intervention): Study subjects will continue their current antiretroviral regimens, which include a protease inhibitor or efavirenz plus two nucleoside analog reverse-transcriptase inhibitors (NRTIs).
- Raltegravir arm. (Experimental): Study subjects will switch their protease inhibitor or efavirenz to once daily raltegravir plus continue current nucleoside analog reverse-transcriptase inhibitors (NRTIs).
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — The aim of this study is to investigate whether switching a protease inhibitor (PI) or efavirenz to raltegravir has effect on liver fat and metabolism in HIV-infected patients who are overweight or obese and have at least one metabolic syndrome component .
  Other Names: Isentress
  Arms: Raltegravir arm.

SUMMARY:
This study will provide data on the switch from a protease inhibitor or efavirenz to the new formulation of raltegravir (RAL) dosed once daily. The study group consists of patients with metabolic risk factors and co-morbidities, in need of optimization of their current ART to minimize the drug-related metabolic side effects as standard of care.

The primary objective of this study is to investigate whether switching a protease inhibitor (PI) or efavirenz to raltegravir once daily reduces liver fat in patients who are overweight or obese and have at least one metabolic syndrome component. For this purpose, the liver fat content will be analyzed using the proton magnetic resonance spectroscopy.

In addition, the aim is to clarify the change in the body composition and metabolism in this study group. For this purpose the visceral adipose tissue (VAT) and subcutaneous adipose tissue (SAT) volumes will be measured and subcutaneous tissue samples will be collected for future analyses of adipose tissue function.

DETAILED DESCRIPTION:
The prevalences of overweight (body-mass-index, BMI 25-30 kg/m2) and obesity (BMI>30 kg/m2) are steadily increasing among HIV-infected patients globally. In parallel, the risk of non-alcoholic fatty liver disease (NAFLD) increases. Clinically alarming are the data which suggest that HIV infected have higher rates of progressive form of NAFLD than non-HIV infected age, gender and BMI matched controls.

As the treatment for HIV is life-long, it is crucial to understand the effects of different antiretroviral therapy (ART) regimens on metabolism. Some antiretroviral agents appear to promote unfavourable changes in metabolism (e.g. in blood lipids) and predispose to trunk fat redistribution and liver fat accumulation.

Raltegravir has been demonstrated to have beneficial impact on some metabolic parameters compared to the protease inhibitor class or efavirenz. In this study, the aim is to investigate whether switching a protease inhibitor or efavirenz to raltegravir reduces liver fat in patients who are overweight or obese and have at least one metabolic syndrome component. For this purpose, the proton magnetic resonance spectroscopy will be used.

In addition, the aim is to clarify the change in the body composition in this study group. For this purpose, the visceral adipose tissue (VAT) and subcutaneous adipose tissue (SAT) volumes will be measured using MRI.

To acquire more knowledge on metabolic effects in adipose tissue level, subcutaneous adipose tissue biopsies will be collected together with blood, saliva and feces samples.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* HIV-positive adult (age over 18) subjects currently on stable ART, with no changes in the ART regimens during the past 6 months.
* Current ART includes either a protease inhibitor or efavirenz.
* No documented or suspected resistance to integrase inhibitors or to NRTIs.
* No prior history of virologic failure. Failure is defined as a confirmed plasma viral load > 200 cop/ml measured no less than six months after initiation or modification of therapy.
* Virological blips accepted only if a single viral load measurement has been between 50-200 cop/ml followed by viral load < 50 cop/ml without the need to initiate a change in ART and no blip within 12 month window period prior to screening.
* Documented evidence of at least two HIV viral load < 50 cop/ml measurements during the past 12 months prior to inclusion: one within 6 months prior to screening.
* HIV viral load < 50 cop/ml at screening.
* BMI>25 kg/m2 and one metabolic syndrome condition, which are

  * BP ≥ 130/≥ 85 mmHg or hypertension medication currently in use or
  * fasting glucose ≥ 5.6 mmol/l or B-HbA1C > 42 mmol/mol or diabetes medication currently in use or
  * HDL < 1.0 mmol/l in men and < 1.3 mmol/l in women or triglycerides ≥ 1.7 mmol/l or a cholesterol-lowering regimen currently in use or
  * waist circumference > 94 cm in men and >80 cm in women (or respective cut off values for non-European ethnic groups as defined by International Diabetes Federation). OR
* ultrasound or biopsy proven hepatosteatosis.

Exclusion Criteria:

* Within 12 month window period prior to screening, HIV viral load measurement of >50 cop/ml.
* More than one consecutive HIV viral load measurements of > 50 cop/ml in the treatment history after initial viral suppression with ART.
* Chronic hepatitis B or C.
* Daily alcohol consumption ≥ 30 g for men and ≥ 20 g for women.
* Pregnancy or planned pregnancy during the study period.
* Lipid or glucose lowering regimen or hormonal supplement started within 3 months before the planned study start.
* Psychiatric disorder, which prevents a study subject to understand the study protocol.
* Other serious disease, which prevents a study subject to participate in the study.
* For MRI/spectroscopy imaging: metal objects in the body or claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Sutinen, MD PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Aurora hospital, Department of Infectious Diseases, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanttu AM, Pekkala S, Satokari R, Hartikainen AK, Arkkila P, Pietilainen KH, Sutinen JP. Gut microbiota alterations after switching from a protease inhibitor or efavirenz to raltegravir in a randomized, controlled study. AIDS. 2023 Feb 1;37(2):323-332. doi: 10.1097/QAD.0000000000003419. Epub 2022 Nov 10. PMID 36541643
- [Derived] Hanttu A, Vuoti S, Kivela P, Arkkila P, Lundbom N, Hakkarainen A, Lundbom J, Lehtimaki T, Viskari H, Lehtinen V, Pietilainen KH, Sutinen J. Liver Fat, Adipose Tissue, and Body Composition Changes After Switching from a Protease Inhibitor or Efavirenz to Raltegravir. AIDS Patient Care STDS. 2021 Sep;35(9):335-341. doi: 10.1089/apc.2021.0106. PMID 34524919

RESULTS

PARTICIPANT FLOW:
Groups:
- Control (= no Intervention Arm).: Study subjects will continue their current antiretroviral regimens, which include a protease inhibitor or efavirenz plus two nucleoside analog reverse-transcriptase inhibitors (NRTIs).
Period: Overall Study
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm.
Started | 24 | 21
Completed | 24 | 19
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm. | Total
Number analyzed (Participants) | 24 | 19 | 43
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [43 to 62] | 49 [39 to 54] | 49 [42 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 19 | 15 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 22 | 18 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Finland | 24 | 19 | 43
Liver fat content [Median (Inter-Quartile Range); unit: % hepatic fat fraction] — %, measured by proton magnetic resonance spectroscopy Population: Only those participants with data available at the specified time points were analyzed.
  % hepatic fat fraction
    number analyzed (Participants) | 23 | 19 | 42
    (all) | 3.1 [1.6 to 7.3] | 2.3 [1.1 to 6.0] | 2.3 [1.4 to 5.8]
Subcutaneous adipose tissue volume [Median (Inter-Quartile Range); unit: mL] — Population: Only those participants with data available at the specified time points were analyzed.
  mL
    number analyzed (Participants) | 22 | 18 | 40
    (all) | 5377 [3693 to 8237] | 3979 [2068 to 6468] | 4468 [2547 to 6146]
Visceral adipose tissue volume [Median (Inter-Quartile Range); unit: mL] — Population: Only those participants with data available at the specified time points were analyzed.
  mL
    number analyzed (Participants) | 22 | 18 | 40
    (all) | 2053 [1906 to 2886] | 1795 [1249 to 3164] | 1906 [1539 to 2349]
Body weight [Median (Inter-Quartile Range); unit: kg] — Population: Only those participants with data available at the specified time points were analyzed.
  kg
    number analyzed (Participants) | 23 | 19 | 42
    (all) | 98.8 [89.2 to 106.7] | 85.9 [76.1 to 97.7] | 93.2 [80.4 to 101.1]
Total body fat [Median (Inter-Quartile Range); unit: kg] — Measured by bioelectrical impedance analysis. Population: Only those participants with data available at the specified data points were analyzed.
  kg
    number analyzed (Participants) | 23 | 19 | 42
    (all) | 30.0 [23.6 to 48.6] | 20.3 [14.6 to 29.7] | 23.8 [17.3 to 32.5]
Liver stiffness [Median (Inter-Quartile Range); unit: kPa] — Measured by transient elastography (Fibroscsan). Population: Only those participants with data available at the specified time points were analyzed.
  kPa
    number analyzed (Participants) | 22 | 19 | 41
    (all) | 4.7 [4.1 to 5.5] | 4.1 [3.3 to 5.6] | 4.4 [3.6 to 5.5]
Fasting plasma glucose [Median (Inter-Quartile Range); unit: mmol/L] — Population: Only those participants with data available at the specified time points were analyzed.
  mmol/L
    number analyzed (Participants) | 23 | 19 | 42
    (all) | 6.0 [5.7 to 6.3] | 5.5 [5.3 to 6.0] | 5.7 [5.5 to 6.3]
Fasting serum LDL cholesterol [Median (Inter-Quartile Range); unit: mmol/L] — Population: Only those participants with data available at the specific data points were analyzed.
  mmol/L
    number analyzed (Participants) | 22 | 19 | 41
    (all) | 3.2 [2.8 to 3.5] | 3.2 [2.7 to 3.6] | 3.2 [2.7 to 3.5]
Fasting serum HDL cholesterol [Median (Inter-Quartile Range); unit: mmol/L] — Population: Only those participants with data available at the specified data points were analyzed.
  mmol/L
    number analyzed (Participants) | 23 | 19 | 42
    (all) | 1.13 [0.98 to 1.28] | 1.30 [1.02 to 1.39] | 1.20 [1.01 to 1.39]
Fasting serum triglyceride [Median (Inter-Quartile Range); unit: mmol/L] — Population: Only those participants with data available at the specified data points were analyzed.
  mmol/L
    number analyzed (Participants) | 23 | 19 | 42
    (all) | 1.3 [1.1 to 1.8] | 1.3 [1.1 to 2.2] | 1.3 [1.1 to 1.8]
Serum high sensitivity CRP [Median (Inter-Quartile Range); unit: mg/L] — Population: Only those participants with data available at the specified data points were analyzed.
  mg/L
    number analyzed (Participants) | 23 | 19 | 42
    (all) | 2.4 [1.0 to 3.7] | 1.0 [0.6 to 2.4] | 1.3 [0.7 to 2.7]
Serum IL-6 [Median (Inter-Quartile Range); unit: pg/mL] — Population: Only those participants with data available at the specified data points were analyzed.
  pg/mL
    number analyzed (Participants) | 22 | 19 | 41
    (all) | 2.2 [2.0 to 4.0] | 2.4 [1.5 to 3.3] | 2.2 [1.7 to 3.1]

OUTCOME MEASURES:

1. Primary Outcome: Change in Liver Fat
Description: 24 week value minus baseline value, liver fat % measured by proton magnetic resonance spectroscopy.
Time Frame: Baseline and 24 weeks
Population: Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: % hepatic fat fraction
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm.
Number analyzed (Participants) | 21 | 18
% hepatic fat fraction | 0.3 [-0.5 to 2.7] | 0.6 [-0.3 to 1.6]

2. Secondary Outcome: Change in Subcutaneous and Visceral Adipose Tissue Volume
Description: 24 week value minus baseline value: change in subcutaneous (SAT) and visceral (VAT) adipose tissue volume (mL) measured by magnetic resonance imaging. Analysis included a series of T1-weighted trans-axial images from 8 cm above to 8 cm below the 4th and 5th lumbar intervertebral disc (16 slices, field of view 375 x 500 mm2, slice thickness 10 mm).
Time Frame: Baseline and 24 weeks
Population: Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm.
Number analyzed (Participants) | 21 | 18
mL
  Change in SAT (24 weeks - baseline) | -74 [-627 to 202] | 242 [27 to 341]
  Change in VAT (24 weeks - baseline) | 100 [-126 to 569] | 66 [-149 to 299]

3. Secondary Outcome: Change in Body Weight and Total Body Fat
Description: 24 week value minus baseline value, change in body weight (kg) and total body fat (kg) measured by Bioelectrical Impedance Analysis.
Time Frame: Baseline and 24 weeks
Population: Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm.
Number analyzed (Participants) | 21 | 18
kg
  Change in body weight (24 weeks - baseline) | 0.9 [-1.8 to 4.1] | 2.0 [0.4 to 3.3]
  Change in body fat (24 weeks - baseline): number analyzed (Participants) | 21 | 17
  Change in body fat (24 weeks - baseline) | -0.3 [-1.7 to 1.5] | 1.5 [0.1 to 2.5]

4. Other Pre Specified Outcome: Change in Liver Stiffness
Description: 24 week minus baseline value, change in liver stiffness (kPa) measured by transient elastography (Fibroscan ®).
Time Frame: Baseline and 24 weeks
Population: Only those participants with data available at the specified data points were analyzed.
Measure: Median (Inter-Quartile Range); unit: kPa
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm.
Number analyzed (Participants) | 19 | 18
kPa | -0.5 [-1.2 to 0.6] | -0.2 [-1.6 to 0.9]

5. Other Pre Specified Outcome: Change in Fasting Plasma Glucose
Description: 24 week value minus baseline value, change in fasting plasma glucose (mg/dL).
Time Frame: Baseline and 24 weeks
Population: Only those participants with data available at the specified data points were analyzed.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm.
Number analyzed (Participants) | 21 | 17
mg/dL | 0.0 [-7.2 to 5.4] | -1.8 [-10.8 to 0.0]

6. Other Pre Specified Outcome: Change in Fasting Serum Lipid Profile
Description: 24 week value minus baseline value, change in fasting serum lipid profile: LDL and HDL cholesterol, triglyceride (all values in mmol/L)
Time Frame: Baseline and 24 weeks
Population: Only those participants with data available at the specified data points were analyzed.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm.
Number analyzed (Participants) | 20 | 18
mmol/L
  Change in fasting serum LDL (24 weeks - baseline) | 0.1 [-0.4 to 0.4] | -0.5 [-1.0 to -0.1]
  Change in fasting serum HDL (24 weeks - baseline) | 0.04 [-0.07 to 0.15] | -0.07 [-0.16 to -0.01]
  Change in fasting serum triglycerides (24 weeks - baseline) | -0.05 [-0.28 to 0.20] | -0.18 [-0.49 to 0.19]

7. Other Pre Specified Outcome: Change in Metabolic and Inflammatory Biomarkers: hsCRP
Description: 24 week value minus baseline value, change in circulating metabolic and inflammatory biomarkers: high sensitivity C-reactive protein (hsCRP mg/L)
Time Frame: Baseline and 24 weeks
Population: Only those participants with data available at the specified data points were analyzed.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm.
Number analyzed (Participants) | 20 | 17
mg/L | 0.66 [-0.07 to 1.45] | -0.06 [-0.59 to 0.22]

8. Other Pre Specified Outcome: Change in Metabolic and Inflammatory Biomarkers: IL-6
Description: 24 week value minus baseline value, change in circulating metabolic and inflammatory biomarkers: interleukin 6 (IL-6 pg/mL)
Time Frame: Baseline and 24 weeks
Population: Only those participants with data available at the specified data points were analyzed.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm.
Number analyzed (Participants) | 20 | 17
pg/mL | 0.83 [-0.09 to 1.20] | 0.00 [-0.87 to 0.64]

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Control (= no Intervention Arm). | Raltegravir Arm.
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/19
Other Adverse Events (participants affected / at risk) | 20/24 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (= no Intervention Arm). (N=24) | Raltegravir Arm. (N=19)
Acute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (= no Intervention Arm). (N=24) | Raltegravir Arm. (N=19)
Headache (Nervous system disorders) | 8 | 9
Gastrointestinal (diarrhoea, nausea) (Gastrointestinal disorders) | 7 | 9
Sleeping difficulties (Psychiatric disorders) | 13 | 10
Nervousness (Psychiatric disorders) | 9 | 7
Dizzyness (Nervous system disorders) | 8 | 5
Depressed mood (Psychiatric disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT03374358/Prot_SAP_000.pdf